CLINICAL TRIAL: NCT02286284
Title: Usefulness of Extracorporeal Removal of sFlt-1 in Women With Severe Preeclampsia at Less Than 26 Weeks' Gestation
Brief Title: Usefulness of Extracorporeal Removal of sFLT-1 in Women With Very Early Severe Preeclampsia
Acronym: ADENA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety of patients : CSI recommandation and promotor decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130928/ N°IDRCB2014-A01044-43
Record Dates: First submitted 2014-11-03; First posted 2014-11-07 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-06

CONDITIONS: Preeclampsia
Keywords: Early severe preeclampsia; Angiogenic factor; Apheresis
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apheresis arm (Experimental): Apheresis for extracorporal removal of sFlt-1
  Interventions: Device: Apheresis for extracorporal removal of sFlt-1

INTERVENTIONS:
Device: Apheresis for extracorporal removal of sFlt-1

SUMMARY:
Introduction Preeclampsia is a multifactorial disease that is responsible of important adverse maternal and perinatal outcomes. Recently, it has been suggested that soluble fms-like tyrosine kinase 1, s-Flt1, induces preeclampsia-like phenotype in experimental models and circulates at elevated levels in human preeclampsia.

The aim of our study is to see whether removal of s-Flt1 may improve perinatal death in women with very early severe preeclampsia at less than 26 weeks' gestation Patients and methods Phase II trial. Women with singleton pregnancy having severe preeclampsia at 23-256/7 weeks' gestation. Women under 18 years, with multiples, or severe fetal growth restriction (less than 5th centile), or abnormal fetal heart rate, or maternal complications (abruption, eclampsia, HELLP syndrome, pulmonary edema, DIC, liver hematoma) are excluded from the study. After blood pressure and maternal stabilization, women are approached for information and if they agree, to sign the trial consent.

Women have twice weekly extracorporeal removal of s-Flt1 until 34 weeks' gestation.

Primary endpoint or success of the procedure: baby alive or alive at 6 months if hospitalized Statistical procedure Simon minimax plan; P0: 60%, P1, 90%, alpha error: 5%, beta power; 90%. First step: number 8 patients. If success equal or less than 5, the study is stopped.

Second step: if success of 6 or more, the study is continued for 9 more patients.

Overall, a maximum of 17 patients will be included. The final success of extracorporeal removal of s-Flt1 will be considered if 14 or more babies will be alive or alive at 6 months if hospitalized.

DETAILED DESCRIPTION:
Introduction Preeclampsia is a multifactorial disease that is responsible of important adverse maternal and perinatal outcomes. Recently, it has been suggested that soluble fms-like tyrosine kinase 1, s-Flt1, induces preeclampsia-like phenotype in experimental models and circulates at elevated levels in human preeclampsia.

The aim of our study is to see whether removal of s-Flt1 may improve perinatal death in women with very early severe preeclampsia at less than 26 weeks' gestation Patients and methods Phase II trial. Women with singleton pregnancy having severe preeclampsia at 23-256/7 weeks' gestation. Women under 18 years, with multiples, or severe fetal growth restriction (less than 5th centile), or abnormal fetal heart rate, or maternal complications (abruption, eclampsia, HELLP syndrome, pulmonary edema, DIC, liver hematoma) are excluded from the study. After blood pressure and maternal stabilization, women are approached for information and if they agree, to sign the trial consent.

They will then be admitted to the department of Renal intensive care of Tenon Hospital. LDL apheresis will be performed twice weekly, during 90 minutes per session, using the DALI 750 Kit and the ART device (Fresenius). sFlt1 will be measured in peripheral blood before and after each session. The treatment will end when delivery is indicated (whether because of threatening complications or because a viable term of pregnancy is achieved).

Primary endpoint or success of the procedure: a live born baby alive at 6 month after birth.

Secondary endpoints: days of pregnancy prolongation, blood pressure during apheresis, fetal heart rate monitoring after apheresis, maternal levels of s-Flt1, PlGF, and s-endoglin.

Maternal adverse outcomes: eclampsia, HELLP syndrome, DIC, pulmonary edema, abruption placentae, renal failure.

Neonatal outcome: gestational age at delivery, birth weight, Apgar score, patent ductus arteriosus, RDS, PVL, IVH, NEC, days in NICU.

Statistical procedure Simon minimax plan; P0: 60%, P1, 90%, alpha error: 5%, beta power; 90%. First step: number 8 patients. If success equal or less than 5, the study is stopped.

Second step: if success of 6 or more, the study is continued for 9 more patients.

Overall, a maximum of 17 patients will be included. The final success of extracorporeal removal of s-Flt1 will be considered if 14 or more babies will be alive at 6 months after birth

ELIGIBILITY:
Inclusion Criteria:

* Severe preeclampsia at less than 26 weeks' gestation
* Singleton pregnancy
* Signed consent

Exclusion Criteria:

* Multiple pregnancy
* Gestational age at 26 or above weeks' gestation
* Estimated foetal weight at diagnosis <5th percentile
* Abnormal fetal heart rate at entry, where feasible (>24 weeks' gestation)
* Maternal complications at diagnosis: Uncontrolled blood pressure, HELLP syndrome, abruption, eclampsia pulmonary edema, renal failure, liver hematoma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Baby discharged alive or alive at 6 months if hospitalized | 6 months
  During the first step (inclusion of 8 patients) analysis is done continuously, and if 3 women have unsuccess primary endpoint, first step and the study are stopped, with a conclusion of failure of the procedure of lipapheresis.

SECONDARY OUTCOMES:
Pregnancy prolongation and preeclampsia related adverse outcomes | 15 weeks
  The data will be measured during the participation of the patient : 15 weeks = 11 weeks of pregnancy monitoring (from 23 to 34 weeks' gestation) + 4 weeks postpartum
Immunoadsorption tolerance for the mother during the session of lipapheresis | 11 weeks
  A description of the following variables will be used: blood pressure during the session, infectious or hemorrhagic events subsequent infusion and / or technique. The time frame is 11 weeks as a maximum : 11 weeks of pregnancy monitoring (from 23 to 34 weeks' gestation)
Foetal immunoadsorption tolerance during the session of lipapheresis | 11 weeks
  Measuring of the heart monitoring's data will be used. The time frame is 11 weeks as a maximum : 11 weeks of pregnancy monitoring (from 23 to 34 weeks' gestation)
Circulating levels of sFlt1, the placental growth factor (PlGF) and soluble endoglin (sEng) until deliverance | 12 weeks
  For the measure of the maternal adsorptive efficiency, the following parameters will be described: circulating levels of sFlt1, the placental growth factor (PlGF) and soluble endoglin (sEng). The time frame is 12 weeks : 11 weeks of pregnancy monitoring (from 23 to 34 weeks' gestation) + until deliverance

CONTACTS AND LOCATIONS:
Overall Officials: Bassam HADDAD, Principal Investigator — CHIC Creteil
Locations (1):
- CHIC, Créteil, France

REFERENCES:
- [Background] Anedda S, Mura S, Marcello C, Pintus P. HELP LDL-apheresis in two cases of familial hypercholesterolemic pregnant women. Transfus Apher Sci. 2011 Feb;44(1):21-4. doi: 10.1016/j.transci.2010.12.004. Epub 2011 Jan 22. PMID 21257349
- [Background] Belghiti J, Kayem G, Tsatsaris V, Goffinet F, Sibai BM, Haddad B. Benefits and risks of expectant management of severe preeclampsia at less than 26 weeks gestation: the impact of gestational age and severe fetal growth restriction. Am J Obstet Gynecol. 2011 Nov;205(5):465.e1-6. doi: 10.1016/j.ajog.2011.06.062. Epub 2011 Jun 24. PMID 21889120
- [Background] Cashin-Hemphill L, Noone M, Abbott JF, Waksmonski CA, Lees RS. Low-density lipoprotein apheresis therapy during pregnancy. Am J Cardiol. 2000 Nov 15;86(10):1160, A10. doi: 10.1016/s0002-9149(00)01183-8. PMID 11074223
- [Background] Deis S, Rouzier R, Kayem G, Masson C, Haddad B. Development of a nomogram to predict occurrence of preeclampsia. Eur J Obstet Gynecol Reprod Biol. 2008 Apr;137(2):146-51. doi: 10.1016/j.ejogrb.2007.05.022. Epub 2007 Jul 31. PMID 17669579
- [Background] Azizi M, Chedid A, Oudard S. Home blood-pressure monitoring in patients receiving sunitinib. N Engl J Med. 2008 Jan 3;358(1):95-7. doi: 10.1056/NEJMc072330. No abstract available. PMID 18172185
- [Background] Chelbi ST, Veitia RA, Vaiman D. Why preeclampsia still exists? Med Hypotheses. 2013 Aug;81(2):259-63. doi: 10.1016/j.mehy.2013.04.034. Epub 2013 May 10. PMID 23669375
- [Background] Eremina V, Sood M, Haigh J, Nagy A, Lajoie G, Ferrara N, Gerber HP, Kikkawa Y, Miner JH, Quaggin SE. Glomerular-specific alterations of VEGF-A expression lead to distinct congenital and acquired renal diseases. J Clin Invest. 2003 Mar;111(5):707-16. doi: 10.1172/JCI17423. PMID 12618525
- [Background] Haddad B, Masson C, Deis S, Touboul C, Kayem G; College national des gynecologues et obstetriciens; Societe francaise de medecine perinatale; Societe francaise de neonatalogie; Societe francaise de anesthesie et de reanimation. [Criteria of pregnancy termination in women with preeclampsia]. Ann Fr Anesth Reanim. 2010 Apr;29(4):e59-68. doi: 10.1016/j.annfar.2010.02.019. Epub 2010 Mar 27. French. PMID 20347561
- [Background] Haddad B, Deis S, Goffinet F, Paniel BJ, Cabrol D, Siba BM. Maternal and perinatal outcomes during expectant management of 239 severe preeclamptic women between 24 and 33 weeks' gestation. Am J Obstet Gynecol. 2004 Jun;190(6):1590-5; discussion 1595-7. doi: 10.1016/j.ajog.2004.03.050. PMID 15284743
- [Background] Kabbinavar F, Hurwitz HI, Fehrenbacher L, Meropol NJ, Novotny WF, Lieberman G, Griffing S, Bergsland E. Phase II, randomized trial comparing bevacizumab plus fluorouracil (FU)/leucovorin (LV) with FU/LV alone in patients with metastatic colorectal cancer. J Clin Oncol. 2003 Jan 1;21(1):60-5. doi: 10.1200/JCO.2003.10.066. PMID 12506171
- [Background] Levine RJ, Qian C, Maynard SE, Yu KF, Epstein FH, Karumanchi SA. Serum sFlt1 concentration during preeclampsia and mid trimester blood pressure in healthy nulliparous women. Am J Obstet Gynecol. 2006 Apr;194(4):1034-41. doi: 10.1016/j.ajog.2005.10.192. PMID 16580293
- [Background] Maynard SE, Min JY, Merchan J, Lim KH, Li J, Mondal S, Libermann TA, Morgan JP, Sellke FW, Stillman IE, Epstein FH, Sukhatme VP, Karumanchi SA. Excess placental soluble fms-like tyrosine kinase 1 (sFlt1) may contribute to endothelial dysfunction, hypertension, and proteinuria in preeclampsia. J Clin Invest. 2003 Mar;111(5):649-58. doi: 10.1172/JCI17189. PMID 12618519
- [Background] Romero R, Nien JK, Espinoza J, Todem D, Fu W, Chung H, Kusanovic JP, Gotsch F, Erez O, Mazaki-Tovi S, Gomez R, Edwin S, Chaiworapongsa T, Levine RJ, Karumanchi SA. A longitudinal study of angiogenic (placental growth factor) and anti-angiogenic (soluble endoglin and soluble vascular endothelial growth factor receptor-1) factors in normal pregnancy and patients destined to develop preeclampsia and deliver a small for gestational age neonate. J Matern Fetal Neonatal Med. 2008 Jan;21(1):9-23. doi: 10.1080/14767050701830480. PMID 18175241
- [Background] Steegers EA, von Dadelszen P, Duvekot JJ, Pijnenborg R. Pre-eclampsia. Lancet. 2010 Aug 21;376(9741):631-44. doi: 10.1016/S0140-6736(10)60279-6. Epub 2010 Jul 2. PMID 20598363
- [Background] Sugimoto H, Hamano Y, Charytan D, Cosgrove D, Kieran M, Sudhakar A, Kalluri R. Neutralization of circulating vascular endothelial growth factor (VEGF) by anti-VEGF antibodies and soluble VEGF receptor 1 (sFlt-1) induces proteinuria. J Biol Chem. 2003 Apr 11;278(15):12605-8. doi: 10.1074/jbc.C300012200. Epub 2003 Jan 21. PMID 12538598
- [Background] Thadhani R, Kisner T, Hagmann H, Bossung V, Noack S, Schaarschmidt W, Jank A, Kribs A, Cornely OA, Kreyssig C, Hemphill L, Rigby AC, Khedkar S, Lindner TH, Mallmann P, Stepan H, Karumanchi SA, Benzing T. Pilot study of extracorporeal removal of soluble fms-like tyrosine kinase 1 in preeclampsia. Circulation. 2011 Aug 23;124(8):940-50. doi: 10.1161/CIRCULATIONAHA.111.034793. Epub 2011 Aug 1. PMID 21810665
- [Background] Thadhani R, Mutter WP, Wolf M, Levine RJ, Taylor RN, Sukhatme VP, Ecker J, Karumanchi SA. First trimester placental growth factor and soluble fms-like tyrosine kinase 1 and risk for preeclampsia. J Clin Endocrinol Metab. 2004 Feb;89(2):770-5. doi: 10.1210/jc.2003-031244. PMID 14764795